CLINICAL TRIAL: NCT04602156
Title: Randomized Comparison of US-guided TROcar Versus SELdiger Technique for Percutaneous Cholecystostomy. The TROSELC II Trial.
Brief Title: US-guided Trocar Versus Seldiger Technique for Percutaneous Cholecystostomy
Acronym: TROSELCII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Stavros Spiliopoulos, Assistant Professor in Interventional Radiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EBD 515/16-9-2020
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Cholecystitis
Keywords: Percutaneous cholecystostomy; ultrasound-guided; interventional radiology; Trocar; Seldinger
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (Experimental): Patients will be randomized to undergo PC catheter placement (8-French) using the trocar method under US guidance while receiving local anesthesia and opioid analgesic, in a bedside setting, either in the US room or in the ICU.
  Interventions: Procedure: Trocar percutaneous cholecystostomy
- Group S (Active Comparator): Patients will be randomized to undergo PC catheter placement (8-French) using the Sellinger method under US guidance while receiving local anesthesia and opioid analgesic, in a bedside setting, either in the US room or in the ICU.
  Interventions: Procedure: Seldinger percutaneous cholecystostomy

INTERVENTIONS:
Procedure: Trocar percutaneous cholecystostomy — Percutaneous cholecystostomy using the one-step Trocar technique under US guidance. An 8Fr Trocar catheter will be inserted percutaneously within the gallbladder under real-time US guidance. The procedure will be performed using an aseptic technique, local anesthesia and intravenous opioid analgesia.
  Arms: Group T
Procedure: Seldinger percutaneous cholecystostomy — Percutaneous cholecystostomy using the Seldinger technique under US guidance. Following percutaneous puncture of the gallbladder with an 18G needle under real-time US guidance, an 8Fr catheter will be inserted percutaneously over the wire within the gallbladder under real-time US guidance. The procedure will be performed using an aseptic technique, local anesthesia and intravenous opioid analgesia.
  Arms: Group S

SUMMARY:
A single-center randomized comparison of bedside ultrasound (US)-guided trocar technique versus the US-guided Seldinger technique for percutaneous cholecystostomy

DETAILED DESCRIPTION:
This is a single-center, randomized, controlled trial (RCT), comparing bedside US-guided trocar technique versus the US-guided Seldinger technique for percutaneous cholecystostomy (PC). The study will randomize a total of 100 consecutive patients (50 in each group) undergoing PC at one large tertiary university hospital. The primary endpoints will be technical success and procedure-related complication rates. Secondary endpoints will be procedural duration, pain assessment, and clinical success after up to 3 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring PC, regardless of the underlying cause.
* Signed informed consent form

Exclusion Criteria:

* Age <18 years or >100 years
* The necessity for CT-guided PC catheter placement, according to the judgment of the performing physician
* Severe uncontrollable coagulopathy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Technical success | At the end of the procedure
  Image verified catheter placement within the gallbladder and subsequent bile aspiration
Procedure-related complications | 3 months
  Minor or major complications attributed to the procedure

SECONDARY OUTCOMES:
Duration of the procedure | Intraprocedural
  The time period between administration of local anesthesia and pigtail catheter positioning within the gallbladder
Intraprocedural pain | End of the procedure
  pain experienced during the procedure assessed using a standard visual analogue score the procedure, as assessed using a standard visual analog score
Post-procedural pain | 12 hours
  Pain experienced up to12 hours after procedure assessed using a standard visual analogue score (VAS - Visual Analog Scale 0-10, 0 representing no pain & 10 representing worst pain experienced)
Clinical success | 72 hours
  Gradual subsidence of signs, symptoms, and elevated inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Spiliopoulos, MD, PhD, Principal Investigator — ATTIKO University Hospital
Locations (1):
- "Attikon" University General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
IPD could be available upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD could be available after the completion of the study upon reasonable request
Access Criteria: email